CLINICAL TRIAL: NCT03734276
Title: Effect of High-intensity Training on the Level of Physical Activity After Thoracoscopy Surgery: a Pilot Study
Acronym: HITAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haute Ecole de Santé Vaud (Other)
Responsible Party: Sponsor
Organization: HEDSV (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERVD 2018-01511
Record Dates: First submitted 2018-10-29; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Rehabilitation; Thoracic Surgery; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: feasibility Study with randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity exercise (Experimental)
  Interventions: Other: High intensity activity
- Control (Active Comparator)
  Interventions: Other: control arm

INTERVENTIONS:
Other: High intensity activity — Cyclo-ergometer session in high intensity setting
  Arms: High intensity exercise
Other: control arm — Usual care
  Arms: Control

SUMMARY:
Goal of this study is to evaluate management with high intensity re-entrainment during the postoperative hospital phase.

This type of early treatment with as little intervention time has so far never been done. The investigators therefore want to carry out this feasibility study in order to collect the data needed to calculate the number of randomized control trial. Investigators will also evaluate the feasibility of this project concerning recruitment, intervention in the hospital phase and data collection once the return home. The evaluation of the activity will be done one month after the return to home by means of a actigraphy of one week.

ELIGIBILITY:
Inclusion Criteria:

* Indication of thoracoscopic surgery
* Autonomous mobilization (with or without auxiliary device)

Exclusion Criteria:

* Patient dependent on oxygen before the procedure
* chronic obstructive pulmonary disease patient with forced expiratory volume at one second <50% predicted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of the intervention on the level of physical activity when returning home by actigraphy | change from baseline number of steps at 7 days after back home and at 30 days after back home
  Number of steps per day during 5 days

SECONDARY OUTCOMES:
Evaluate the impact of the intervention on the level of physical activity by questionnaires. | change from baseline questionnaire at 7 days after back home and at 30 days after back home
  "Inventaire du Soi Physique - 6" questionnaire
Evaluate the impact of the intervention on the level of physical activity by questionnaires. | change from baseline questionnaire at 7 days after back home and at 30 days after back home
  "International Physical Activity Questionnaire-- Short Form

IPD SHARING:
Plan to Share IPD: Undecided